CLINICAL TRIAL: NCT05782881
Title: High Risk Population of Cardiovascular Disease in Hubei Province (Coronary Heart Disease With Diabetes) Screening and Intervention Program
Brief Title: High Risk Population of Cardiovascular Disease in Hubei Province Screening and Intervention Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCDInT
Record Dates: First submitted 2023-02-18; First posted 2023-03-24 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Cardiovascular Diseases; Diabetes Mellitus, Type 2; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2; Coronary Disease | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Angiotensin-Converting Enzyme Inhibitors; Glucagon-Like Peptide 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protocol treatment group (Experimental): Strictly intervene blood glucose, blood pressure and blood lipids
  Interventions: Behavioral: phone calls and encouraging patients' lifestyle change and medication adherence; Drug: Statin
- Conventional treatment group (Placebo Comparator): Treatment and management according to the guidelines
  Interventions: Drug: Statin

INTERVENTIONS:
Behavioral: phone calls and encouraging patients' lifestyle change and medication adherence — Use some methods to strictly intervene blood glucose , blood pressure and blood lipids for protocol treatment group people.
  Arms: Protocol treatment group
Drug: Statin — Treatment and management according to the guidelines
  Other Names: Angiotensin-converting enzyme inhibitor; Angiotensin receptor neprilysin inhibitor; Glucagon-like peptide-1; Sodium-dependent glucose transporters 2

SUMMARY:
High Risk Population of Cardiovascular Disease in Hubei Province (Coronary Heart Disease With Diabetes) Screening and Intervention Program（CCDInT）is a randomized controlled study to verify that protocol treatment group is more effective than the conventional treatment group in reducing the incidence of composite cardiovascular disease (cardiovascular death, non fatal myocardial infarction, non fatal stroke, hospitalization for heart failure, and readmission for acute coronary syndrome) in patients with coronary heart disease and type 2 diabetes.

DETAILED DESCRIPTION:
The overall objective of the High Risk Population of Cardiovascular Disease in Hubei Province (Coronary Heart Disease With Diabetes) Screening and Intervention Program（CCDInT） will be carried out in medical institutions in 14 prefecture level cities (prefectures) in Hubei province that could meet the test requirements. A total of 16,000 individuals aged ≥40 years with coronary heart disease with diabetes will be recruited into the study. Study participants will be followed in 1 year for some study outcomes. The main purpose of this study is to verify that the protocol treatment group is more effective than the conventional treatment group in reducing the incidence of composite cardiovascular disease (cardiovascular death, non fatal myocardial infarction, non fatal stroke, hospitalization for heart failure, and readmission for acute coronary syndrome) in patients with coronary heart disease and type 2 diabetes. In addition, the investigators will further study the genetic mechanism of compound cardiovascular events from the molecular genetic level, and explore the contribution and impact of genetic diversity on the treatment effect. At the same time, explore and establish a cardiovascular disease prevention and control system and effective mechanism under the leadership of provincial and municipal health administrative departments, organized by provincial prevention and control centers, and guided by municipal and state prevention and control centers, which provide theoretical and experimental basis for formulating strategies for large-scale intervention of related diseases, so as to improve the prevention and control status and effect, and strive to reduce the disease and social burden.

ELIGIBILITY:
Inclusion Criteria:

1. 40-75 years old, male or female
2. Patients with coronary heart disease complicated with type 2 diabetes (confirmed by angiography)
3. Low density lipoprotein cholesterol >1.8mmol/l
4. Willing to participate and sign informed consent

Exclusion Criteria:

1. Received coronary stent treatment in recent one year
2. Pregnant or lactating women
3. Decompensated stage of chronic systolic heart failure (NYHA cardiac function rating ≥ 3), cardiac function; Patients with severe cardiovascular complications such as septic shock
4. Stroke patients in recent 1 year
5. Patients with severe gastrointestinal diseases, liver failure or kidney failure
6. Cancer patients or patients who have received radiotherapy or chemotherapy within five years
7. Suffering from infectious diseases such as AIDS and tuberculosis
8. Hospitalized or suffering from other serious diseases requiring immediate hospitalization
9. Bad addicts: drug users or alcoholics (men >80 g / day, women >40 g / day)
10. Disturbance of consciousness, inability to communicate normally or any mental illness; Those who are inconvenient to take care of themselves or move
11. Life expectancy <12 months
12. Individuals with abnormal laboratory tests and clinical manifestations who are judged by the researcher to be unsuitable for participation
13. Unwilling to participate in the trial, unwilling to change the current drug treatment plan

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16000 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite cardiovascular disease (cardiovascular death, non fatal myocardial infarction, non fatal stroke, hospitalization for heart failure, and readmission for acute coronary syndrome) | 1 year after baseline
  Record the composite cardiovascular disease(cardiovascular death, non fatal myocardial infarction, non fatal stroke, hospitalization for heart failure, and readmission for acute coronary syndrome)

SECONDARY OUTCOMES:
All-cause death | 1 year after baseline
  Number of all-cause death
All-cause mortality | 1 year after baseline
  Record all-cause mortality
Cardiovascular death | 1 year after baseline
  Record cardiovascular death
non-fatal myocardial infarction | 1 year after baseline
  Record non-fatal myocardial infarction
non-fatal stroke | 1 year after baseline
  Record non-fatal stroke
readmission for heart failure | 1 year after baseline
  Record readmission for heart failure
readmission for acute coronary syndrome | 1 year after baseline
  Number of patients with readmission for acute coronary syndrome
Diabetic nephropathy | 1 year after baseline
  Number of patients with Diabetic nephropathy
Proportion of hypertension control (BP<140/90 mm Hg) | 1 year after baseline
  Record proportion of hypertension control (BP<140/90 mm Hg)
Proportion of low density lipoprotein-cholesterol(LDL-C<1.4mmol/L) | 1 year after baseline
  Record proportion of low density lipoprotein-cholesterol(LDL-C<1.4mmol/L)
Proportion of glycosylated hemoglobin(GHb<7.0%) | 1 year after baseline
  Record proportion of glycosylated hemoglobin(GHb<7.0%)
Blood pressure( both diastolic and systolic will be measured) | baseline, 3 months after baseline, 6 months after baseline, 12 months after baseline
  Record blood pressure( both diastolic and systolic will be measured)

CONTACTS AND LOCATIONS:
Overall Officials: Kai Huang, doctor, Study Chair — Union Hospital, Tongji Medical College of Huazhong University of science and technology; Yong Huo, doctor, Study Chair — Peking University First Hospital
Locations (107):
- China (107):
  - Affiliated Minzu University Hospital of Hubei Minzu University, Enshi, Hubei
  - Badong Peolple's Hospital, Enshi, Hubei
  - Enshi Central Hospital, Enshi, Hubei
  - Laifeng People's Hospital, Enshi, Hubei
  - Lichuan People's Hospital, Enshi, Hubei
  - The Central Hospital of Enshi Tujia and Miao Autonomous Prefecture, Enshi, Hubei
  - The People's Hospital of Jianshi, Enshi, Hubei
  - Xianfeng County People's Hospital, Enshi, Hubei
  - Xuanen People's Hospital, Enshi, Hubei
  - Ezhou Central Hospital, Ezhou, Hubei
  - Ezhou Hospital of Chinese Medicine, Ezhou, Hubei
  - Hongan People's Hospital, Huanggang, Hubei
  - Huangmei Peolple's Hospital, Huanggang, Hubei
  - Luotian People's Hospital, Huanggang, Hubei
  - People's Hostpital of Macheng City, Huanggang, Hubei
  - Qichun People's Hospital, Huanggang, Hubei
  - The People's Hospital of Tuanfeng, Huanggang, Hubei
  - Wuxue People's Hopital, Huanggang, Hubei
  - Xishui People's Hospital, Huanggang, Hubei
  - Yingshan People's Hospital, Huanggang, Hubei
  - Daye People's Hospital, Huangshi, Hubei
  - Huangshi Central Hospital, Huangshi, Hubei
  - Huangshi Love&Health Hospital Affiliated of Hubei Polytechnic University, Huangshi, Hubei
  - Yangxin People's Hospital, Huangshi, Hubei
  - Jingmen NO.1 People's Hospital, Jingmen, Hubei
  - Jingmen NO.2 People's Hospital, Jingmen, Hubei
  - Jingshan Union Hospital of Huazhong University of Science and Technology, Jingmen, Hubei
  - Zhongxiang Hospital of Traditional Chinese Medicine, Jingmen, Hubei
  - Zhongxiang People's Hospital, Jingmen, Hubei
  - Chinese Medicine Hospital of Gongan, Jingzhou, Hubei
  - Chinese Medicine Hospital of Honghu, Jingzhou, Hubei
  - Jiangling People's Hospital, Jingzhou, Hubei
  - Jianli Hospital of Chinese Medicine, Jingzhou, Hubei
  - Jianli People's Hospital, Jingzhou, Hubei
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - Jingzhou Hospital of Traditional Chinese Medicine, Jingzhou, Hubei
  - Jingzhou No.1 People's Hospital, Jingzhou, Hubei
  - People's Hospital of Gongan, Jingzhou, Hubei
  - People's Hospital of Honghu, Jingzhou, Hubei
  - Shishou People's Hostpital, Jingzhou, Hubei
  - Songzi of Traditional Chinese Medicine, Jingzhou, Hubei
  - Songzi People's Hospital, Jingzhou, Hubei
  - The Second Hospital of Jingzhou, Jingzhou, Hubei
  - The Second People's Hospital of Jianli, Jingzhou, Hubei
  - Danjiangkou First Hospital, Shiyan, Hubei
  - Fang County People's Hospital, Shiyan, Hubei
  - Shiyan Renmin Hospital, Shiyan, Hubei
  - Sinopharm Dongfeng General Hospital, Hubei University of Medicine, Shiyan, Hubei
  - Taihe Hospital, Shiyan, Hubei
  - Xunyang People's Hospital, Shiyan, Hubei
  - Yunxi People's Hospital, Shiyan, Hubei
  - Zhushan People's Hospital, Shiyan, Hubei
  - Zhuxi Hospital of Traditional Chinese Medicine, Shiyan, Hubei
  - NO.1 Peoples Hospital of Guangshui, Suizhou, Hubei
  - People's Hospital of Suixian, Suizhou, Hubei
  - Suizhou Central Hospital, Suizhou, Hubei
  - Suizhou Hospital of Traditional Chinese Medicine, Suizhou, Hubei
  - Suizhou Zengdu Hospital, Suizhou, Hubei
  - The First People's Hospital of Tianmen in Hubei Province, Tianmen, Hubei
  - CR & WISCO General Hospital, Wuhan, Hubei
  - Fifth Hospital in Wuhan, Wuhan, Hubei
  - Hospital of Universal Love, Wuhan, Hubei
  - People's Hospital of Dongxihu District, Wuhan, Hubei
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - Union Hospital, Tongji Medical College of Huazhong University of science and technology, Wuhan, Hubei
  - Wuhan NO.1 Hospital, Wuhan, Hubei
  - Wuhan Third Hospital-Tongren Hospital of Wuhan University, Wuhan, Hubei
  - Huanggang Central Hospital, Wuhan, Hubei
  - Baokang People's Hospital, Xiangyang, Hubei
  - Gucheng People's Hospital, Xiangyang, Hubei
  - Laohekou NO.1 Hospital, Xiangyang, Hubei
  - Nanzhang People's Hospital, Xiangyang, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Xiangyang Hospital of Traditional Chinese Medicine, Xiangyang, Hubei
  - Xiangyang NO.1 People's Hospital, Xiangyang, Hubei
  - Xiangzhou People's Hospital, Xiangyang, Hubei
  - Yicheng People's Hosptital, Xiangyang, Hubei
  - Zaoyang NO.1 People's Hospital, Xiangyang, Hubei
  - Chibi General Hospital, Xianning, Hubei
  - Chongyang People's Hospital, Xianning, Hubei
  - Jiayu People's Hospital, Xianning, Hubei
  - The First People's Hospital of Xianning, Xianning, Hubei
  - TongchengPeople's Hospital, Xianning, Hubei
  - Tongshan People's Hospital, Xianning, Hubei
  - Xianning Central Hospital, Xianning, Hubei
  - AMHT Hubei Aerospace Hospital, Xiaogan, Hubei
  - Anlu Puai Hospital, Xiaogan, Hubei
  - Dawu County Hosptal of Traditional Chinese Medicine, Xiaogan, Hubei
  - Dawu People's Hospital, Xiaogan, Hubei
  - Hanchuan People's Hospital, Xiaogan, Hubei
  - The Central Hospital of Xiaogan, Xiaogan, Hubei
  - Xiaochang First People's Hospital, Xiaogan, Hubei
  - Xiaogan First People's Hospital, Xiaogan, Hubei
  - Xiaogan Hoospital of Chinese Medicine, Xiaogan, Hubei
  - Yingcheng People's Hospital, Xiaogan, Hubei
  - Yunmeng People's Hospital, Xiaogan, Hubei
  - Affiliated Renhe Hospital of China Three GORGES University, Yichang, Hubei
  - People's Hospital of Dangyang, Yichang, Hubei
  - People's Hospital of Zhijiang, Yichang, Hubei
  - People's Hospital of Zigui, Yichang, Hubei
  - Sinopharm Gezhouba Central Hospital, Yichang, Hubei
  - The First Hospital of YC, Yichang, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - Yichang Hospital of Traditional Chinese Medicine, Yichang, Hubei
  - Yichang Second People's Hospital, Yichang, Hubei
  - Yidu People's Hospital, Yichang, Hubei
  - Yiling Hospital of Yichang, Yichang, Hubei

IPD SHARING:
Plan to Share IPD: No
The overall objective of the High Risk Population of Cardiovascular Disease in Hubei Province (Coronary Heart Disease With Diabetes) Screening and Intervention Program will use Case Report Form scale, and data input and management were carried out by Electronic Data Capture System .